CLINICAL TRIAL: NCT00843336
Title: Randomized Comparison of Two Internet Supported Natural Family Planning Methods
Brief Title: Comparison of Two Internet Supported Natural Family Planning Methods
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Richard J. Fehring, Professor, Marquette University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FPR200801363
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy
Keywords: fertility monitoring; contraception
MeSH Terms: interventions — Long-Term Synaptic Depression; Blood Glucose Self-Monitoring; Ovulation Detection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic hormonal fertility monitoring (Experimental): Use of an electronic hormonal fertility monitor that measures urinary estrogen and LH and provides users with low, high, or peak fertility readings.
  Interventions: Behavioral: Electronic hormonal fertility monitoring
- Cervical mucus monitoring (Active Comparator): Self-monitoring of externally observed cervical mucus to determine level of fertility.
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Electronic hormonal fertility monitoring — Use of an electronic hormonal fertility monitor that provides three levels of fertility; low, high, and peak. Monitor is based upon urinary levels of E3G (estrogen) and LH. Monitor readings are placed in an electronic charting system on the Internet.
  Other Names: ClearBlue Easy Fertility Monitor (Unipath, LTD).
  Arms: Electronic hormonal fertility monitoring
Behavioral: Self-monitoring — Self-monitoring of externally observed cervical mucus to determine level of fertility.
  Other Names: Ovulation method
  Arms: Cervical mucus monitoring

SUMMARY:
The purpose of this research study is to compare the effectiveness of two natural family planning (NFP) methods that are provided over the internet by the Marquette University Institute for Natural Family Planning. One of the NFP methods is the use of a hand held electronic hormonal fertility monitor. The other method involves the self-observation of cervical mucus to track fertility. Both of the methods will involve placing information about fertility into an online charting system that automatically displays the days of fertility and infertility. The investigators are also interested in the influence of mutual motivation by the woman and her partner in using these methods to avoid pregnancy. The investigators hypothesize that there will be lower unintended pregnancy rates among those couples who use the electronic hormonal fertility monitor and among those couples who have a strong motivation to avoid pregnancy.

DETAILED DESCRIPTION:
The Office of Population Affairs (OPA) of the Department of Human Development recently submitted a call for proposals for research on methods of natural family planning (NFP). The department chairs of OPA have recognized that relatively few women in the United States use natural methods of family planning, especially in the Title X Family Planning programs and clinics. They wanted researchers to develop studies to help increase the use and the efficacy of these methods, and, furthermore, wanted to understand why the methods are not used more. Reasons why only about 0.2% of US women use natural methods of birth control are they are often difficult to use, they are relatively ineffective, and there is a lack of access to properly trained NFP teachers. At Marquette University we have developed simple methods of NFP that utilize an electronic fertility monitor that measures female reproductive hormones, self cervical mucus monitoring that estimates the fertile window, and a simple fertility formula to help estimate the beginning and end of the fertile window. We also have developed a Web site that offers easy access to information on NFP, electronic charting, and professional nurses with specialization in teaching NFP.

The specific purpose of our study is to determine the efficacy, satisfaction, ease of use, and motivation in using an internet based NFP method that utilizes an electronic hormonal fertility monitor plus a simple fertility formula (i.e., EHFM-NFP) within an online professional-nurse supported system. Since there are few studies that compare methods of NFP, another aim of this study is to compare an internet based EFHM-NFP method with an internet based traditional cervical mucus monitoring (CMM) NFP method - both methods were developed at Marquette University. Please note that we have 3 published efficacy studies of the Marquette Method.

The specific research questions that will be asked are:

1. What are the 3, 6, and 12-month unintended pregnancy rates of an internet-provided EHFM-aided NFP method?
2. What are the 3, 6, and 12-month unintended pregnancy rates of an internet-provided CMM-only NFP method?
3. What is the satisfaction, ease of use, and mutual motivation of an internet-based NFP method (either EFHM or CMM) over a 12-month time period, i.e., after 1, 3, 6, and 12 months of use?

ELIGIBILITY:
For Female participants

Inclusion Criteria:

* be between the age of 18 and 42
* be in a sexually active committed relationship with a man
* have a menstrual cycle range of 21-42 days

Exclusion Criteria:

* have not used Depo (injectable) contraception for the past 6 months
* have not used oral or patch hormonal contraception for the past 3 months
* have not breast-fed baby for at least three months
* have no known fertility problems
* not be using medications that interfere with fertility
* not smoke cigarettes; and
* not be pregnant.

For Male Participants

Inclusion criteria:

* be between the ages of 18 and 50
* be in a sexually active committed relationship with his lone woman partner.

Exclusion criteria:

* have no known fertility problems

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 358 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Unintended Pregnancies | 1, 3, 6, and 12 months
  Survival analysis of based on unintended pregnancies and correct use menstrual cycles (for perfect use analysis) and typical use (based on total number of menstrual cycles) -- to be calculated at 1, 3, 6, and 12 months of use. A Kaplan-Meier survival curve over that time period will be displayed to show change.

SECONDARY OUTCOMES:
user satisfaction, ease of use, mutual motivation | 1, 3, 6 and 12 months; mutual motivation monthly
  To determine if there is significant change from baseline (at 1 month) to 3, 6 and 12 months in the outcome measure of "satisfaction and ease of use" - repeated measure analysis (ANOVA) will be used. Change in motivation to avoid pregnancy from baseline (i.e., before charting the first menstrual cycle) through 12 months of use will also be analyzed for changes by repeated measure analysis. We will also use repeated measure analysis to determine differences in the outcome measures between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Fehring, PhD, Principal Investigator — Marquette University College of Nursing
Locations (2):
- United States (2):
  - Marquette University College of Nursing, Milwaukee, Wisconsin
  - Marquette University, Milwaukee, Wisconsin

REFERENCES:
- [Background] Fehring RJ, Schneider M, Barron ML. Efficacy of the Marquette Method of natural family planning. MCN Am J Matern Child Nurs. 2008 Nov-Dec;33(6):348-54. doi: 10.1097/01.NMC.0000341254.80426.32. PMID 18997569
- [Background] Fehring RJ, Schneider M, Raviele K, Barron ML. Efficacy of cervical mucus observations plus electronic hormonal fertility monitoring as a method of natural family planning. J Obstet Gynecol Neonatal Nurs. 2007 Mar-Apr;36(2):152-60. doi: 10.1111/j.1552-6909.2007.000129.x. PMID 17371516
- [Background] Fehring RJ, Schneider M, Barron ML, Raviele K. Cohort comparison of two fertility awareness methods of family planning. J Reprod Med. 2009 Mar;54(3):165-70. PMID 19370902
- [Derived] Fehring RJ, Schneider M, Raviele K, Rodriguez D, Pruszynski J. Randomized comparison of two Internet-supported fertility-awareness-based methods of family planning. Contraception. 2013 Jul;88(1):24-30. doi: 10.1016/j.contraception.2012.10.010. Epub 2012 Nov 12. PMID 23153900
- See also: Marquette NFP Institute Research Web page — http://www.marquette.edu/nursing/NFP/Research.shtml